CLINICAL TRIAL: NCT01764516
Title: Arak University of Medical Sciences , Ministry of Health and Education,I.R.Iran
Brief Title: Study on Serum Zinc and Selenium Levels in Epileptic Patients
Status: Completed | Type: Observational
Sponsor: Arak University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Farahani Heidar, faculity of medicine, department of biochemistry, Arak University of Medical Sciences
Other Study IDs: f110@1958; f110@19588 (Other Grant/Funding Number: Grant of Arak Medical Sciences University); f110@19588 (Registry Identifier: MD thesis); f110@19588 (Other: ministry of health and education I.R.Iran)
Record Dates: First submitted 2013-01-05; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Generalized Epileptic
Keywords: zinc; selenium; serum; epilepsy; antioxidants
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: None Retained — Serum were analysis for zinc and selenium
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Zinc level (micro gram per deciliter): In all cases
- Selenium level (micro gram per deciliter): In all cases
- Zinc level in male (micro gram per deciliter)
- Selenium level in male (micro gram per deciliter)
- Zinc level in Female (micro gram per decilitre)
- Selenium level in Female (micro gram per decilitre)

SUMMARY:
This study was carried out with the purpose of evaluating zinc and selenium levels in serum of epileptic patients and compare with normal individuals.

DETAILED DESCRIPTION:
Forty patients aged 18 to 50 years visiting Vali-Asr hospital in Arak, I.R. Iran, who were diagnosed with generalized form of epilepsy by a neurologist for the first time were recruited as cases. The control group (n=40) was selected from healthy individuals, in whom no disease was diagnosed until this study, and were matched to the case group by age, sex, and economical status.

ELIGIBILITY:
Inclusion Criteria:

New generalized and single epileptic cases patients who accept and sign the approval form of ethical committee non smoker, no trauma, no use of selenium supplement, no use of zinc supplement, no use of vitamin A supplement, no use of vitamin D supplement, no Weight loss, no Diarrhea, no addiction, no alcohol consumption, no use of certain medications,

Exclusion Criteria:

presence of above criteria as well as, generalized and single epileptic cases under treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all generalized and single epileptic patiants which were identify for fist time
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Study on Serum Zinc and Selenium Levels in Epileptic Patients | 5 months
  decrement in serum zinc and selenium level

SECONDARY OUTCOMES:
Comparison between the selenium levels by gender in two groups | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidar N Farahani, PhD, Principal Investigator — Department of Biochemistry,Arak medical sciences university
Locations (1):
- Vali-Asr Hospital, Arak, Markazi Province, Iran